CLINICAL TRIAL: NCT06088667
Title: The Effect of Fascial Release on Pain, Range of Motion and Functionality After Arthroscopic Rotator Cuff Repair
Brief Title: Fascial Release After Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Director, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Karabuk University 78
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double-blind study; the patients will not be informed about training group or control group and they will be evaluated and trained at different places and times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial mobilization group (Experimental): In addition to the rehabilitation given to the control group, the fascial release group will be treated with the Graston device to the superficial and deep fascia of the neck and shoulder muscles, biceps and triceps brachii muscles and forearm compartments.
  Interventions: Other: Fascial mobilization group
- Control Group (Experimental): The control group will receive heat application, electrical stimulation and shoulder exercises for 4 weeks.
  Interventions: Other: Fascial mobilization group

INTERVENTIONS:
Other: Fascial mobilization group — In addition to the rehabilitation given to the control group, the fascial release group will be treated with the Graston device to the superficial and deep fascia of the neck and shoulder muscles, biceps and triceps brachii muscles and forearm compartments for 4 weeks.

SUMMARY:
Instrument-assisted soft tissue mobilization (IASTM) is a popular treatment method that can be used for myofascial restriction and fascial release. IASTM is used to reduce pain in the area where the pathology is located, increase range of motion (ROM), improve movement function and provide a mobilizing effect. When the literature was examined, no study was found examining the effectiveness of the IASTM technique, which is known to require less effort and stimulate healing compared to manual interventions, in the rehabilitation period after rotator cuff arthroscopic surgery. Therefore, our study aimed to examine the effects of instrument-assisted fascial mobilization given in addition to conventional rehabilitation on long-term pain, function, joint range of motion, fear of movement, and daily living activities in patients who have passed 4 weeks after rotator cuff arthroscopic surgery and are candidates for rehabilitation.

DETAILED DESCRIPTION:
Rotator cuff (RC) rupture causes shoulder pain, muscle weakness, and decreased shoulder range of motion (ROM). Additionally, fear of movement develops due to shoulder pain, affecting ROM and function. Treatment of RC rupture is initially conservative. In cases where conservative treatment is inadequate, surgical option is preferred. Open, mini-open and arthroscopic repair can be used in surgery. In recent years, arthroscopic repair has been mostly preferred because it causes less pain than other surgical options, has a shorter hospital stay, and does not cause complications. A postoperative rehabilitation program is a crucial component of surgical success. The aim of this program is to reduce pain, increase ROM, and improve patients' functional level and activities of daily living. The postoperative rehabilitation program includes electrophysical agents, manual therapy and exercise.Surgery-related inflammation may restrict fascial tissue. Inflammation changes the mechanical properties of connective tissue, causing adhesions and eventually leading to stiffness. Thus, the slip between fascial surfaces decreases and, accordingly, ROM and function decrease.

Instrument Assisted Soft Tissue Mobilization (IASTM) is used for myofascial restriction and fascial release. IASTM is used to reduce pain in the area where the pathology is located, increase range of motion (ROM), improve movement function and provide a mobilizing effect. However, it is noteworthy that there is a lack of studies examining the long-term effectiveness of fascial mobilization in shoulder pathologies. When the literature was examined, no study was found examining the effectiveness of the IASTM technique, which is known to require less effort and stimulate healing compared to manual interventions, in the rehabilitation period after rotator cuff arthroscopic surgery. Therefore, our study aimed to examine the effects of instrument-assisted fascial mobilization given in addition to conventional rehabilitation on long-term pain, function, range of motion, fear of movement, and daily living activities in patients 4 weeks after rotator cuff arthroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* 4 weeks have passed since arthroscopic rotator cuff repair

Exclusion Criteria:

* cervical discopathy,
* shoulder osteoarthritis
* fracture or tumor of the upper extremity,
* adhesive capsulitis,
* shoulder instability,
* thoracic outlet syndrome and
* patients with neurological or mental problems.
* Non-voluntary patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Pain severity | baseline and 4 weeks post-intervention
  Visuel analog scale will be used to evaluate individuals' shoulder pain level.

SECONDARY OUTCOMES:
Range of motion | baseline and 4 weeks post-intervention
  Joint range of motion will be assessed using a universal goniometer
Kinesiophobia | baseline and 4 weeks post-intervention
  The Tampa Kinesiophobia Scale (TSK) will be used to measure individuals' fear of movement/reinjury.
Functional level | baseline and 4 weeks post-intervention
  The Shoulder Pain and Disability Index (SPADI) will be used to evaluate functional disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Physiotherapy and Rehabilitation Application and Research Center, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pegreffi F, Paladini P, Campi F, Porcellini G. Conservative management of rotator cuff tear. Sports Med Arthrosc Rev. 2011 Dec;19(4):348-53. doi: 10.1097/JSA.0b013e3182148dc6. PMID 22089284
- [Background] Nikolaidou O, Migkou S, Karampalis C. Rehabilitation after Rotator Cuff Repair. Open Orthop J. 2017 Feb 28;11:154-162. doi: 10.2174/1874325001711010154. eCollection 2017. PMID 28400883
- [Result] Coban T, Demirdel E, Yildirim NU, Deveci A. The investigation of acute effects of fascial release technique in patients with arthroscopic rotator cuff repair: A randomized controlled trial. Complement Ther Clin Pract. 2022 Aug;48:101573. doi: 10.1016/j.ctcp.2022.101573. Epub 2022 Mar 21. PMID 35397305